CLINICAL TRIAL: NCT05612516
Title: Assessment of Peroxide Level in Saliva During Teeth Bleaching With 9.5% Hydrogen Peroxide Gel Using a Tray With Reservoir Versus a Tray Without Reservoir. A Randomized Clinical Trial
Brief Title: Peroxide Level in Saliva During Teeth Bleaching Using a Tray With Reservoir Versus a Tray Without Reservoir.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Anas Yousef Mohammad, Master Degree student- Faculty of Dentistry, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CU-2-2022
Record Dates: First submitted 2022-11-03; First posted 2022-11-10 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Consumption
Keywords: Home bleaching; Tray with reservoir; Tray without reservoir

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydrogen peroxide 9.5% bleaching using a tray with reservoir. (Active Comparator): . Alginate impressions of maxillary dental arches of patients will be taken to obtain casts and produce the customized trays.
  Reservoirs 1.5 mm thick will be created on the facial surfaces of anterior teeth, including the first premolars in the arches, applying a light-cured resin on the casts. The resin layer thickness will be standardized using a thickness gauge (1.5 mm thickness). Then, customized trays will be fabricated with 1.5 mm-thick vinyl acetate sheets using the thermoforming process. Trays will be precisely trimmed completely involving tooth surface (1.5 mm incisal or occlusal to gingival margin), and the adaptation will be verified on the casts. The trays will be placed over teeth to verify the adaptation in the patients' mouth.
  Interventions: Procedure: Assessment of hydrogen peroxide levels in saliva using trays with reservoir.
- Hydrogen peroxide 9.5% bleaching using a tray without reservoir. (Active Comparator): Alginate impressions of maxillary dental arches of patients will be taken to obtain casts to produce the customized trays. Then, customized trays will be fabricated with no space for reservoir, with 0.9 mm-thick vinyl acetate sheets using the thermoforming process applying a light-cured resin on the casts. Trays will be precisely trimmed completely involving tooth surface (1 mm incisal or occlusal to gingival margin), and the adaptation will be verified on the casts. The trays will be placed over teeth to verify the adaptation in the participants' mouths.
  Interventions: Procedure: Assessment of hydrogen peroxide levels in saliva using trays without reservoir.

INTERVENTIONS:
Procedure: Assessment of hydrogen peroxide levels in saliva using trays with reservoir. — During bleaching using trays with reservoir.
  Arms: Hydrogen peroxide 9.5% bleaching using a tray with reservoir.
Procedure: Assessment of hydrogen peroxide levels in saliva using trays without reservoir. — During bleaching using trays without reservoir.
  Arms: Hydrogen peroxide 9.5% bleaching using a tray without reservoir.

SUMMARY:
The aim of the study is to clinically assess the peroxide levels in saliva during bleaching with 9.5% hydrogen peroxide using a tray with or without reservoir.

DETAILED DESCRIPTION:
Statement of the Problem There is more concern about the possible adverse effect of bleaching agent, patients report gastrointestinal mucosal irritation e.g. a burning palate, throat and minor upsets in the stomach and intestine. Some adverse effects of hydrogen peroxide as a dental bleaching agent include dentin sensitivity and/or gingival irritation led by unstable and reactive H+ free radicals and low pH from prolonged use. Peroxide is a highly reactive substance which can damage oral soft tissues and hard tissues when present in high concentrations and with exposures of prolonged duration. (Alqahtani, 2014). Several researches have focused on the problem of gel ingestion and potential peroxide release in saliva (Dahl et al, 2003; Watt et al, 2004; Bernardon et al, 2010; Goldberg et al, 2010).

Rationale

Reservoirs are modifications in the tray molds to increase the amount of bleaching material carried by the bleaching tray, seeking greater bleaching efficacy. The use of reservoirs in the bleaching trays was initially seen as positive, since higher accumulation of material could provide the patient with greater treatment efficacy. Martini et al, 2020 stated that there is no significant difference between groups whitened with and without reservoirs for gingival irritation or tooth sensitivity. Most authors and bleaching gel manufacturers recommend the use of reservoirs to increase the amount of product available for bleaching and to allow for complete seating of the bleaching tray, although that the reservoirs decrease tray retention and increase lab fabrication time and cost (Javaheri et al, 2000). The presence of reservoirs decreases the retention of the tray, allowing more room for the gel but also reducing the adaptation of the tray. That may cause more leakage of the material, which may lead to more peroxide level in saliva. (Haywood et al, 1992).

A major concern for clinicians was the potential toxicological effect of hydrogen peroxide contacting soft tissues. A safe hydrogen peroxide exposure level (no observed effect level) was determined with catalase-deficient mice, reporting a maximum dose of 26 mg/kg/d. This corresponds to the dose level in humans, considering the conventional uncertainty factor of 100-fold, of 0.26 mg/kg/d (IGHRC, 2003; Hannig et al, 2005; Li et al, 2011). The safety of hydrogen peroxide products used for at home bleaching regarding peroxide release in saliva has not been fully proven.

ELIGIBILITY:
Inclusion Criteria:

1. Good general health.
2. Absence of non-carious cervical lesions, active caries, gingival recession, or periodontal disease.
3. Do not use orthodontics appliance or removable prosthesis.
4. Maxillary anterior teeth without caries, restorations and/or endodontic treatment.
5. Mild generalized staining.

Exclusion Criteria:

1. Smoking or alcohol dependent patients.
2. Pregnancy and lactating women.
3. Parafunctional habits or pathologies.
4. Periapical alterations.
5. Use of medicaments that alter salivary flow.
6. Patients who had already undergone tooth bleaching
7. Patients with severe internal tooth discoloration as tetracycline stain, fluorosis or endodontic treatment.
8. Tooth hypersensitivity.
9. Presence of cracks or fractures.
10. Periodontal affection sign and symptoms.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2024-01-10 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2024-05-08 (Actual)

PRIMARY OUTCOMES:
Hydrogen peroxide level in saliva | 1 min after beginning of the bleaching procedure and application of the tray.
  A spectrophotometry method based on the reaction of 4-aminoantipyrine and phenol with hydrogen peroxide will be adopted. This method will allow the oxidation of peroxide by peroxidase enzyme, resulting in solution color change from transparent to pink. The amount of hydrogen peroxide in saliva will be quantified by an analytic spectrophotometer, which will relate light absorbance with peroxide concentration of each sample.
Hydrogen peroxide level in saliva | 5 min after tray application
  A spectrophotometry method based on the reaction of 4-aminoantipyrine and phenol with hydrogen peroxide will be adopted. This method will allow the oxidation of peroxide by peroxidase enzyme, resulting in solution color change from transparent to pink. The amount of hydrogen peroxide in saliva will be quantified by an analytic spectrophotometer, which will relate light absorbance with peroxide concentration of each sample.
Hydrogen peroxide level in saliva | T2: 10 min after tray application
  A spectrophotometry method based on the reaction of 4-aminoantipyrine and phenol with hydrogen peroxide will be adopted. This method will allow the oxidation of peroxide by peroxidase enzyme, resulting in solution color change from transparent to pink. The amount of hydrogen peroxide in saliva will be quantified by an analytic spectrophotometer, which will relate light absorbance with peroxide concentration of each sample.
Hydrogen peroxide level in saliva | T3: 30 min after tray application
  A spectrophotometry method based on the reaction of 4-aminoantipyrine and phenol with hydrogen peroxide will be adopted. This method will allow the oxidation of peroxide by peroxidase enzyme, resulting in solution color change from transparent to pink. The amount of hydrogen peroxide in saliva will be quantified by an analytic spectrophotometer, which will relate light absorbance with peroxide concentration of each sample.

CONTACTS AND LOCATIONS:
Overall Officials: Iman I ElSayad, Professor, Study Director — Cairo University
Locations (1):
- Faculty of dentistry, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No